CLINICAL TRIAL: NCT06236152
Title: Role of Low Dose Steroids vs Placebo in Addition to Anti-tuberculosis Treatment (ATT) in Regression of Lymph Node Sizes in Patients With Tuberculous Lymphadenopathy
Brief Title: Steroids vs Placebo in Treatment of Tuberculous Lymphadenitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fahad Javed Awan (Other)
Responsible Party: Sponsor-Investigator, Fahad Javed Awan, Doctor, Pak Emirates Military Hospital
Organization: Pak Emirates Military Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PakEmiratesMH1023Fahad
Record Dates: First submitted 2023-12-26; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Tuberculous Lymphadenitis, Cervical
Keywords: Painful cervical lymphadenopathy; Tuberculosis; Tuberculous Lymphadenitis
MeSH Terms: conditions — Tuberculosis, Lymph Node; Tuberculosis | interventions — ferrous sulfate; 1-(2-fluoroethyl)-2-nitroimidazole; Methylprednisolone; Prednisone

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two groups, A and B using lottery method. Group A is receiving the standard of care treatment for tuberculosis plus steroids in a low dose (10 mg per day) whereas Group B is receiving the standard of care plus a placebo
Who Masked: Participant
Masking Description: A single blind study protocol was followed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deltacortil (Active Comparator): Deltacortil 10mg was given in oral formulation once daily for 4 to 6 weeks
  Interventions: Drug: Deltacortril
- Placebo (Placebo Comparator): Iron 150mg was given in oral formulation once daily for 4 to 6 weeks
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate — Ferrous Sulphate was given once daily for 4 to 6 weeks to the patients instead of deltacortil.
  Other Names: Fenim; Fersul
  Arms: Placebo
Drug: Deltacortril — Deltacortil 10mg was given orally once daily for 4 to 6 weeks
  Other Names: Prednisone; Dilacort
  Arms: Deltacortil

SUMMARY:
This study will be conducted as a single blinded randomized control trial. The goal of this clinical trial is to learn about the role of low dose steroids in the resolution of tuberculous lymphadenitis. The prime questions, this clinical trial aims to answer are:

* Is there any role of starting low dose steroids in resolution of lymph node size along side standard anti-tubercular drugs in patients of tuberculous lymphadenitis?
* Do low dose steroid therapy in addition to standard anti-TB drugs prevents or reduces the incidence of complications?

Patients presenting to the out patient department of Pak Emirates Military Hospital, Rawalpindi with tuberculous lymphadenitis will be recruited in the study after a written informed consent. Initial size of two largest lymph nodes will be measured. They will be randomized into two groups, only one of which will be receiving the low dose steroids.

The patients will be followed up on a monthly basis and regression in the lymph node size, if any will be measured. The two groups will be compared at the end of the trial.

DETAILED DESCRIPTION:
Tuberculosis earliest records date back to the origin of civilization itself and yet still it remains one of the most elusive of the diseases still haunting the human population in the third world. Newer dugs and treatment protocols are still remain a major focus of discussion in the academic circles. Pakistan accounts for around 60% of the cases of tuberculosis in the East Mediterranean with an overall prevalence reaching 376 cases per 100,000 population. With such a high prevalence of the disease, it becomes punitive that robust TB control programs are run with an aim of not only rooting out the problem but also scientifically studying it so as to add useful information to the current literature available on the disease. This Randomized Control Trial is being conducted in the Pak-Emirates Military Hospital Rawalpindi, Pakistan which is a tertiary care hospital draining a vast area of the Punjab province of Pakistan since July, 2022 with a single blind study protocol. 140 patients with Tuberculous lymphadenitis of any site were recruited in the study after informed consent from 1st July 2022 till 30th June 2023. Patients were randomly assigned to two groups, A and B using lottery method. Group A is receiving the standard of care treatment for tuberculosis plus steroids in a low dose (10 mg per day) whereas Group B is receiving the standard of care plus a placebo. The regression of the size of lymph nodes is being recorded on a monthly follow up till completion of a 6 month standard Anti-tubercular treatment regimen. The data will be entered in the Statistical Package for Social Sciences version 23.00 at end of the trial and will be analyzed so as to compare the regression of the lymph node size between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with tuberculosis having painful tuberculous lymphadenopathy

Exclusion Criteria:

1. Patients with no tuberculous lymphadenopathy.
2. Patients who are already under treatment for tuberculosis.
3. Patient who developed complications due to anti-TB treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Regression of size of cervical lymph nodes was measured using ultrasound neck | 4 to 5 weeks
  Ultrasound neck was done to measure the sizes of lymph nodes in the patients with tuberculous cervical lymphadenitis at the time of enrollment and then after 6 weeks to see the regression in the sizes of the cervical lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Fahad J Awan, MBBS, Principal Investigator — Pak Emirates Military Hospital; Muhammad Uneeb Ullah, MBBS, Principal Investigator — Pak Emirates Military Hospital
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No